CLINICAL TRIAL: NCT00943319
Title: A Phase I-II Study of Busulfan-fludarabine Conditioning and T-cell Depleted Allogeneic Stem Cell Transplantation for Patients With Advanced Hematologic Malignancies
Brief Title: Busulfan-fludarabine Conditioning and T-cell Depleted Allogeneic Stem Cell Transplantation for Patients With Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0132
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Leukemia; Lymphoma; Myeloma
Keywords: Cancers of the blood
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms, Plasma Cell | interventions — Busulfan; fludarabine; Alemtuzumab; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan and fludarabine (Experimental): Intravenous busulfan (Busulfan®) in combination with fludarabine
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Campath; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Busulfan — Daily intravenous dosing to target AVC
Drug: Fludarabine — Fludarabine dosing will be based on actual body weight. Fludarabine will be infused over 30 minutes before busulfan treatment dose.
Drug: Campath — All patients will receive premedication for Campath (daily doses of 20 mg are repeated for up to five times).
Procedure: Stem Cell Transplant — Infusion of bone marrow and donors(related/ unrelated).

SUMMARY:
The purpose of this study is:

1. To establish the maximally tolerated dose (MTD) of intravenous busulfan (Busulfan®) in combination with fludarabine as conditioning regimen for transplantation with in-vivo T-cell depletion.
2. To evaluate disease free and overall survival after this conditioning regimen in patients with advanced acute myeloid leukemia (AML) and myelodysplastic syndromes (MDS).
3. To evaluate potential pharmacogenomic determinants of toxicity of this regimen.
4. To evaluate potential pharmacogenomic determinants of efficacy of this regimen.

ELIGIBILITY:
Inclusion Criteria:

Phase I portion:

* Relapsed or refractory acute myelogenous or lymphoid leukemia.
* Chronic myelogenous leukemia in accelerated phase or blast-crisis.
* Recurrent or refractory malignant lymphoma or Hodgkin's disease
* Recurrent or refractory multiple myeloma.
* Chronic lymphocytic leukemia, relapsed or with poor prognostic features.
* Myeloproliferative disorder (polycythemia vera, myelofibrosis) with transformation
* Myelodysplastic syndromes with more than 5% blasts.

Phase II portion:

* AML with active disease or beyond CR2.
* MDS with more than 5% blasts.

Exclusion Criteria:

* Clinical progression. Such patients may be treated on other treatment protocols or at the investigator's discretion. Such patients will continue to be monitored for survival and, may be asked to continue to provide specimens for studies of minimal residual disease and immune reconstitution as other treatments are recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Artz, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] O'Donnell PH, Artz AS, Undevia SD, Pai RK, Del Cerro P, Horowitz S, Godley LA, Hart J, Innocenti F, Larson RA, Odenike OM, Stock W, Van Besien K. Phase I study of dose-escalated busulfan with fludarabine and alemtuzumab as conditioning for allogeneic hematopoietic stem cell transplant: reduced clearance at high doses and occurrence of late sinusoidal obstruction syndrome/veno-occlusive disease. Leuk Lymphoma. 2010 Dec;51(12):2240-9. doi: 10.3109/10428194.2010.520773. Epub 2010 Oct 4. PMID 20919852

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Busulfan and Fludarabine
Started | 50
Completed | 49
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Busulfan and Fludarabine
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 39
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: Maximally tolerated area under the curve of intravenous busulfan (Busulfan®) in combination with fludarabine as conditioning regimen for transplantation with in-vivo T-cell depletion. The number reported will be an Area Under the Curve (AUC) measure reported in µmol-min/L.
Time Frame: 5 years
Population: The 36 patients refer to the phase I portion of the study only.
Measure: Number; unit: mmol-min/L
Arm/Group | Busulfan and Fludarabine
Number analyzed (Participants) | 36
mmol-min/L | 6800

2. Secondary Outcome: Overall Survival
Description: Overall Survival measured as median survival in days
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Busulfan and Fludarabine
Number analyzed (Participants) | 50
days | 161 [121 to 305]
Statistical Analysis 1: Comparison: Busulfan and Fludarabine; Test type: Other; Product limit survival estimate; Median Survival time = 161, 95% CI 2-sided [121 to 305]

3. Secondary Outcome: Disease Free Survival
Description: Disease Free Survival measured by median survival time in days
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Busulfan and Fludarabine
Number analyzed (Participants) | 50
days | 172 [85 to 436]
Statistical Analysis 1: Comparison: Busulfan and Fludarabine; Estimated median survival time; Test type: Other; Median Disease Free Survival Time = 172, 95% CI 2-sided [85 to 436]

ADVERSE EVENTS:
Time Frame: 10 years
Arm/Group | Busulfan and Fludarabine
All-Cause Mortality (participants affected / at risk) | 45/49
Serious Adverse Events (participants affected / at risk) | 1/49
Other Adverse Events (participants affected / at risk) | 1/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan and Fludarabine (N=49)
Sepsis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan and Fludarabine (N=49)
Mental Status change (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT00943319/Prot_SAP_000.pdf